CLINICAL TRIAL: NCT03355482
Title: MRI Evaluation Assessing Synovitis to Address the Unmet Need for Reliable Endpoints in SLE
Acronym: MEASURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment, funding
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-09; BMS IM101-636 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus Arthritis
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Depomedrol arm (Active Comparator): Patients are treated with new or ascending doses of subcutaneous methotrexate, and receive a single intramuscular dose of Depomedrol (160mg) at baseline.
  Interventions: Drug: Methylprednisolone
- Placebo arm (Sham Comparator): Patients are treated with new or ascending doses methotrexate, and receive a single intramuscular placebo injection at baseline.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Methylprednisolone — 160mg IM at baseline
  Arms: Depomedrol arm
Drug: Placebos — IM saline injection at baseline
  Arms: Placebo arm

SUMMARY:
This is an exploratory evaluation of MRI as a reliable, sensitive, and accurate outcome measure for clinical trials in SLE arthritis. Forty patients with SLE and moderate to severe synovitis (minimum of 3 tender and 3 swollen joints in wrists and hands) will be randomized to new or increased methotrexate therapy plus a single injection of Depomedrol or a matched placebo at baseline. Methotrexate will be injected subcutaneously once per week at ascending doses. The study will evaluate a range of outcomes discernable by MRI at 3 months and 6 months after baseline. We will also compare MRI findings, clinical endpoints, and biomarker changes in patients that were treated with Depomedrol vs. matched placebo at baseline.

DETAILED DESCRIPTION:
This will be a six month, double blind, randomized, placebo- controlled trial of subcutaneous methotrexate vs methotrexate plus baseline Depomedrol in patients with SLE and >/= 3 tender and 3 swollen joints in the hands and wrists. Patients who are already taking methotrexate </= 15 mg/week may qualify and will have a >/= 2.5 mg/week dose increase at baseline, receiving subcutaneous dosing whether on oral or sc dosing prior to entry. Those not taking methotrexate at baseline will initiate open label treatment in ascending doses beginning at 15 mg/week. All patients will increase methotrexate weekly up to 25 mg as tolerated or until resolution of arthritis. Decreases are allowed as needed.

After randomization, patients may choose to stop or continue any NSAIDs, hydroxychloroquine, or up to 10 mg prednisone if these were being used at screening. All other lupus-specific treatments or medications will be withdrawn. Optimization of methotrexate dose must be completed by Month 2. If additional immune- suppressive medications or steroids become necessary during the trial, patients remain evaluable for the primary endpoint, which is defined by clinical response regardless of treatment. In secondary analyses of Depomedrol vs. placebo, patients treated with rescue interventions will be censored when comparing changes in mean/median synovitis, osteitis RAMRIS or tendinitis scores in the two treatment groups, and they will be included as non- responders in dichotomous endpoints (SRI-4, BICLA). These analyses will also provide useful data for many of the other endpoints (comparisons of MRI vs joint counts and other measures which are valid regardless of treatment). Thus, although off protocol medications will not be encouraged, they will not require removal from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting 4 1997 revised ACR classification criteria or SLICC criteria for SLE.
2. Have active polyarticular arthritis with a minimum of 3 tender and 3 swollen joints or tendons in the hands and wrists observed at the screening visit and a history consistent with BILAG 2004 "B" arthritis.
3. Willing and able to receive weekly subcutaneous methotrexate and intramuscular steroid injections (or placebo injection) as per the protocol.
4. Willing and able to stop current immunosuppressants.
5. Willing and able to undergo MRI and other study procedures (including no known allergy to contrast material).
6. Women of childbearing potential must have a negative pregnancy test at screening and baseline and be willing to use effective contraception after the screening visit until three months after the end of the study.
7. People of any sex or gender 18 to 70 years of age.

Exclusion Criteria:

1. Target Disease Exceptions: Patients with acute nephritis requiring induction therapy, CNS lupus (except chorea, cranial neuropathy, and resolving optic neuritis) or any lupus condition requiring cyclophosphamide, biologics, or IV steroids >/= 500 mg.
2. Medical History and Concurrent Diseases:

   1. Patients incapable of understanding or completing study-related assessments.
   2. Patients with any condition, whether or not related to SLE, which, in the opinion of the investigator, might place a patient at unacceptable risk for participation in the study.
   3. Patients with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ.
   4. Patients who, in the opinion of the investigator, currently abuse drugs or alcohol.
   5. Patients with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
   6. Patients who have received any live vaccines within 2 months of the anticipated first dose of study medication.
   7. Patients with any serious bacterial infection within the last 2 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
   8. Patients at risk for tuberculosis (TB). Patients with active TB within 3 years, even if treated; history of active TB > 3 years ago, unless documented prior anti-TB treatment appropriate in duration and type; current known or suspected active TB; and latent TB not successfully treated (≥ 4 weeks at baseline).
3. Physical and Laboratory Test Findings:

   1. Patients must not be known to be positive for hepatitis B surface antigen.
   2. Patients who are known to be positive for hepatitis C antibody may participate if the presence of hepatitis C virus can be excluded by polymerase chain reaction or recombinant immunoblot assay at screening.
   3. Acute hemolytic anemia with hemoglobin < 7.0 g/dL or known change in Hg by 2.0 g/dL within the last two months unless due to SLE and stable for the past month
   4. WBC < 1500/mm3 (< 1.5 x 109/L) unless due to chronic lupus activity and stable for at least one month
   5. Platelets < 40,000/mm3 (< 3 x 109/L) (If less than 100,000 must have been stable (within a range of 10,000/mm3) either by historical testing of known chronic thrombocytopenic patients within two months of screening or in two tests during the screening period at least one week apart.
   6. Serum creatinine > 2 times the ULN or estimated glomerular filtration rate (eGFR) <40 mL/min/1.73 m2
   7. Serum ALT or AST > 2.5 times the ULN. If currently on methotrexate, patients may repeat this test during the screening period or later rescreen.
   8. Any other laboratory test results that, in the opinion of the investigator, might place a patient at unacceptable risk for participation in the study.
4. Allergies and Adverse Drug Reactions: Known allergy or a history, in the opinion of the investigator or patient, of an unacceptable adverse sensitivity to gadolinium, methotrexate or unacceptable difficulties tolerating intramuscular or subcutaneous injections. Patients may elect lower doses of Depomedrol (1/2 or ¼ the dose) however if there is concern about tolerability of the large dose injection.
5. Prohibited Treatments and/or Therapies:

   1. Patients who have received treatment with an investigational biologic within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose.
   2. Patients who have received cyclophosphamide within 3 months of the Day 1 dose or bolus parenteral steroids >/= 500 mg within 1 month of screening.
   3. Use of rituximab within 6 months prior to Day 1; if > 6 months have elapsed since last rituximab dose, reconstitution of total peripheral B cell counts to predosing range should be documented. If there were no predose levels obtained then B cell counts must be minimally 200 x 106/l which characterizes most SLE patients (Odendahl et al. J Immunol 2000;165:5970-5979).
   4. Ongoing treatment (after the baseline visit) with immune suppressants (such as azathioprine, mycophenolate mofetil, leflunomide, calcineurin inhibitors or belimumab). These may be stopped or tapered as soon as informed consent procedures have been completed at the screening visit.
   5. Prednisone > 20 mg po qd (or equivalent) at the time of the screening visit or > 10 mg po qd (or equivalent) at or after randomization (steroids will additionally be tapered during the study if tolerated). Hydroxychloroquine is not exclusionary if the investigator or patient is unwilling to stop it, but taper will also be encouraged if the patient improves. NSAIDS are not exclusionary, but patients will be asked not to take them on the morning of each monthly visit, until the visit is concluded.
6. Other Exclusion Criteria:

   1. Prisoners or patients who are involuntarily incarcerated.
   2. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
   3. Known contraindication or intolerance or risk of MRI procedures (e.g. permanent pacemakers, cardioverter-defibrillators, other implanted electronic devices, aneurysm clips and other metal implants, procedure-limiting claustrophobia (unless mitigated by the circumstances of the testing MRI for small joints) and severe renal impairment (estimated GFR < 40 mL/min/1.73 m2).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
combined MRI synovitis, osteitis and tendinitis score at 3 months compared to baseline in clinical responders | 3 months
  the sum of the MRI synovitis, osteitis and tendinitis scores at 3 months will be compared to baseline by paired t test for those patients with a clinical response to the treatment regimen (defined as>/= 50% decrease in tender and swollen joints and disease severity scored as BILAG C or D at the 3 month visit). Each MRI parameter will be scored semi-quantitatively according to the OMERACT RA-MRI scoring system (RAMRIS) on a scale of 0-3, with 0=normal, 1=mild, 2=moderate, 3=severe involvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Access Health, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided